CLINICAL TRIAL: NCT06851455
Title: Advancing Skills and Confidence in Ultrasound-Guided Injection Techniques: the Impact of a Cadaveric Workshop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Collaborators: Saglik Bilimleri Universitesi (Other); Koç University (Other)
Responsible Party: Principal Investigator, Mert Zure, Ass. Prof. Mert Zure, Saglik Bilimleri Universitesi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: University of Health Sciences
Record Dates: First submitted 2025-02-22; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Ultrasound-Guided Injection; Joint Diseases; Cadaveric Training
Keywords: Ultrasound-guided injection; Cadaveric training; Musculoskeletal ultrasonography; Medical education
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cadaveric Workshop Participants (Experimental): The arm is participant physicians for the workshop that are working in the department of physical medicine and rehabilitation. They are from different academic degrees such as residents, specialists and professors.
  Interventions: Other: Cadaveric Workshop on Ultrasound-guided Injections

INTERVENTIONS:
Other: Cadaveric Workshop on Ultrasound-guided Injections — Participant physicians will attend a structured cadaveric workshop on ultrasound-guided musculoskeletal injections.
  Participants will perform hands-on procedures under expert supervision on lower extremity joints listed as hip, knee and ankle.
  For the assessment participants will be asked to complete pre- and post-workshop assessments to measure skill improvement and confidence levels.

SUMMARY:
The goal of this study is to assess whether a cadaveric ultrasound-guided injection workshop improves procedural skills and confidence among participant physicians. It will also evaluate participants' satisfaction and perceived clinical applicability.

The main questions it aims to answer are:

Does the workshop enhance participants' accuracy and confidence in performing ultrasound-guided musculoskeletal injections? How do participants rate the workshop's effectiveness in improving their clinical skills?

Participants will:

Attend a structured cadaveric workshop on ultrasound-guided musculoskeletal injections.

Perform hands-on procedures under expert supervision. Complete pre- and post-workshop assessments to measure skill improvement and confidence levels.

DETAILED DESCRIPTION:
Ultrasound-guided musculoskeletal injections have become an essential skill in physical medicine and rehabilitation, orthopedic practice, and pain management. Despite their increasing use, mastering these techniques requires both theoretical knowledge and hands-on experience. Cadaveric training workshops provide a unique opportunity for physicians to refine their procedural skills in a controlled environment that closely mimics real-world clinical scenarios.

This study evaluates the effectiveness of a cadaveric musculoskeletal system ultrasound-guided injection workshop in enhancing the technical proficiency, confidence, and clinical readiness of physicians. By integrating structured didactic sessions with hands-on practice on cadaveric specimens, the workshop aims to bridge the gap between theoretical learning and clinical application.

Participants will undergo a comprehensive learning experience, beginning with instructional lectures covering the principles of ultrasound guidance, needle visualization techniques, and common musculoskeletal injection sites. Following this, they will engage in supervised hands-on practice on cadaveric specimens, allowing them to refine their accuracy in needle placement, optimize probe handling, and gain a deeper understanding of anatomical structures.

To assess the workshop's effectiveness, physicians will complete pre- and post-training evaluations, including objective assessments of their procedural accuracy and subjective self-reports on confidence levels. The study will analyze improvements in needle placement precision, injection efficiency, and participants' perceived ability to translate these skills into clinical practice.

By providing an immersive and interactive training experience, this study seeks to determine whether cadaveric workshops serve as a valuable tool in advancing physicians' competency in ultrasound-guided musculoskeletal injections. Findings from this research may contribute to the development of more structured training programs, ultimately improving patient outcomes in musculoskeletal care.

ELIGIBILITY:
Inclusion Criteria:

* Being a physician working in the field of Physical Medicine & Rehabilitation
* Participating in the cadaveric workshop
* Signed the informed consent to participate in the study

Exclusion Criteria:

* Unwilling to provide data for this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2024-10-03 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Pre-Workshop Evaluation Survey | Once at the beginning of the study, just before the workshop
  A pre-workshop survey filled out by participants prior to the lectures, which contained question items about their age, sex, academic and professional experience in medicine and physiatry, prior exposure to MSK USG and injections, current access to ultrasound equipment, prior attendance at other ultrasound training programs, frequency of ultrasound-guided injections done in a week, and self-confidence regarding hip, knee and ankle ultrasound-guided injections using a 5-point Likert scale, with 0 denoting the least confidence and 4 denoting the highest.
Post-Workshop Evaluation Survey | Once, immediately after the workshop
  A post-workshop survey filled out by participants after the workshop to assess their self-confidence in MSK ultrasound-guided injections regarding the three joints and the perceived value of the course. In addition, the usefulness of the course and contentment of participants about the materials used and quality of context were also measured using a 5-point Likert scale, where 0 indicated the least content and 4 the most content. At last, participants were invited to suggest regions, subjects and techniques they would like to have covered in upcoming ultrasonography seminars.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Kanuni Sultan Süleyman Training and Research Hospital, University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided